CLINICAL TRIAL: NCT02335528
Title: SimCoach Evaluation: A Virtual Human Intervention to Encourage Servicemember Help-seeking for PTSD and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-504 W74V8H-06-C-0002; NCT03103165 (obsolete NCT alias)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Post-traumatic Stress Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SimCoach intervention (Experimental): Participants randomized to the SimCoach intervention arm interacted with "Bill Ford," a simulated human (avatar) enacted in the SimCoach program. This white male avatar representing himself as an Army veteran who spoke to participants in a conversational manner. Participants interacted with him using a chat interface, where they could type responses to him. Bill Ford asked participants a series of questions that corresponded to validated PTSD or depression screening questionnaires. SimCoach then provided personalized recommendations for a symptom if the user reported experiencing the symptom at one of the two highest frequencies on the response scale. These recommendations consisted of a behavioral recommendation with an accompanying link to a website or online article on the topic.
  Interventions: Behavioral: SimCoach
- Content Matched Control (No Intervention): Participants assigned to the Content Matched Control condition arm completed text-based versions of the PCL PTSD screening inventory and PHQ-9 depression screening inventory. These instruments used standard, validated language and did not use the modified conversational versions used in the SimCoach intervention condition. The same personalized recommendations provided to the SimCoach group were provided as conventional text and links. After receiving personalized recommendations, participants completed text versions of primary help-seeking, perceived barriers to seeking help, and secondary outcome (user experience) measures.
- No-Treatment Control (No Intervention): Participants randomized to the No-Treatment Control arm completed measures of the primary outcome (intentions to seek help) prior to being given a choice of SimCoach or the conventional screening administered in the other two arms of the study. After the help-seeking intention questionnaire was administered, participants were told that they would be asked some questions about any PTSD or depression symptoms that they might be having and were given the choice between chatting online with a virtual human or using an online form (options were presented in random order to prevent any influence of ordering on selection of the tool). After either interacting with SimCoach or filling out an online form, participants completed a questionnaire assessing user experience.

INTERVENTIONS:
Behavioral: SimCoach
  Arms: SimCoach intervention

SUMMARY:
SimCoach, a computer program featuring a virtual human that speaks and gestures in a videogame-like interface, is designed to encourage servicemembers, especially those with signs or symptoms of post-traumatic stress disorder (PTSD) or depression, to seek help to improve their psychological health. The assessment included a formative component assessing SimCoach's design, development, and implementation approaches, as well as a summative component assessing outcomes among participants in a user experience survey and a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and
* active duty or Reserve servicemember or National Guard servicemember and
* being off duty

Exclusion Criteria:

* under the age of 18 years
* retired servicemember or not a servicemember
* currently on duty
* currently incarcerated, on parole, or on probation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Help-seeking intentions | within 30 days
  Participants were asked the following question: "How likely is it that you will seek help for issues such as stress, emotional, alcohol, drug, or family problems from the following people in the next month?" and responded using a Likert scale ranging from 1=extremely unlikely to 7=extremely likely.
Perceived barriers to care | within 30 days
  Subjects were asked about their perceptions of both stigma-related and practical barriers to seeking help.

SECONDARY OUTCOMES:
User experience | Immediately following their interaction with SimCoach or online form (up to 5 min)
  Participants responded to questions about their experience with the tool or the online form.